CLINICAL TRIAL: NCT03639480
Title: A Double-blind, Randomized, Multi-center Phase 3 Clinical Trial to Evaluate the Safety and Efficacy of CJ-30061 Compared With Amlodipine/Valsartan Combination Therapy and Valsartan/Atorvastatin Combination Therapy in Hypertensive Patients With Hyperlipidemia
Brief Title: Study to Evaluate the Safety and Efficacy of CJ-30061 in Hypertensive Patients With Hyperlipidemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CJ_EXA_301
Record Dates: First submitted 2018-08-09; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Amlodipine; Valsartan; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test (Experimental): Amlodipine 10mg+Valsartan 160mg+Atorvastatin 40mg
  Interventions: Drug: Amlodipine 10mg+Valsartan 160mg+Atorvastatin 40mg
- Reference 1 (Active Comparator): Amlodipine 10mg+Valsartan 160mg
  Interventions: Drug: Amlodipine 10mg+Valsartan 160mg
- Reference 2 (Active Comparator): Valsartan 160mg+Atorvastatin 40mg
  Interventions: Drug: Valsartan 160mg+Atorvastatin 40mg

INTERVENTIONS:
Drug: Amlodipine 10mg+Valsartan 160mg+Atorvastatin 40mg — Amlodipine 10mg+Valsartan 160mg+Atorvastatin 40mg
  Arms: Test
Drug: Amlodipine 10mg+Valsartan 160mg — Amlodipine 10mg+Valsartan 160mg
  Arms: Reference 1
Drug: Valsartan 160mg+Atorvastatin 40mg — Valsartan 160mg+Atorvastatin 40mg
  Arms: Reference 2

SUMMARY:
To evaluate the safety and efficacy of CJ-30061 compared with amlodipine/valsartan combination therapy and valsartan/atorvastatin combination therapy in hypertensive patients with hyperlipidemia

ELIGIBILITY:
Inclusion Criteria:

* Aged between 19 and 74 years
* Diagnosed with essintial hypertension(average siSBP ≥ 140mmHg) accompanying hyperlipidemia(LDL-C ≥ 100mg/dL) and were on or off treatment at Visit 1(screening)
* Decided to participate in the study and provided signed informed consent form voluntarily after receiving explanation of the objectives, methods, and effects of the study

Exclusion Criteria:

* Severe hypertension defined as average siDBP ≥ 120mmHg or average siSBP ≥ 200mmHg at Visit 1(screening)
* The difference in BPs between those measured at the reference arm at Visit 1(screening) was ≥ 10mmHg for siDBP or ≥ 20mmHg for siSBP
* LDL-C > 250mg/dL or TG ≥ 400mg/dL at Visit 1(screening)
* Secondary hypertension
* Diagnosis of type 1 diabetes mellitus(DM) or uncontrolled DM(patients on insulin therapy or patients with HbA1c ≥ 9%)

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-10-13 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Change in siSBP | baseline and 8 weeks
  Change in siSBP from baseline after 8 weeks of study treatment
Change in LDL-C | baseline and 8 weeks
  Change in LDL-C from baseline after 8 weeks of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Duk-Hyun Kang, Ph.D, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea